CLINICAL TRIAL: NCT04091113
Title: Hereditary Angioedema Kininogen Assay: A Multicenter, Epidemiological, Observational Study.
Brief Title: Hereditary Angioedema Kininogen Assay
Acronym: HAEKA
Status: Terminated | Type: Observational
Why Stopped: we will update quickly
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: HAEKA 01-2019
Record Dates: First submitted 2019-09-06; First posted 2019-09-16 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary Angioedema; Cleaved high-molecular weight kininogen; Hereditary Angioedema Type I; Hereditary Angioedema Type II
MeSH Terms: conditions — Angioedemas, Hereditary; Hereditary Angioedema Types I and II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Hereditary Angioedema: Participants older than 18 years that are clinically diagnosed with Hereditary Angioedema type 1/2 and experienced ≥4 HAE attacks within last 12 month before the enrollment

SUMMARY:
A multicenter epidemiological observational study aiming to explore the cleaved high-molecular weight kininogen (cHMWK) including identification and characterization of other metabolite/biomarkers in HAE type 1/2 patients

DETAILED DESCRIPTION:
Hereditary angioedema (HAE) is a rare autosomal dominant genetic disorder characterized by recurrent tissue angioedema episodes, mainly caused by mutations in the SERPING1 gene that encodes C1 inhibitor (C1-INH), a protease involved in limiting bradykinin production. Low levels of C1-INH (HAE type 1) or dysfunctional C1-INH (HAE type 2) lead to bradykinin accumulation, resulting in capillary leakage and tissue swelling.

High Molecular Weight Kininogen (HMWK) proteolysis, by active plasma kallikrein, results in bradykinin and cHMWK generation.

The goal of this study is to explore the cHMWK concentrations in HAE type 1/2 patients, as a biomarker for this disease.

The HAEKA study is performed in collaboration with Shire. Shire is a wholly owned subsidiary of Takeda Pharmaceutical Company Limited.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent is obtained from the participant
* The patient with diagnosis of Hereditary Angioedema (HAE) type 1/2 based on international guidelines
* The patient experienced ≥4 HAE attacks within last 12 month before enrolment in the study
* The participant is older than 18 years old

Exclusion Criteria:

* Inability to provide informed consent
* The patient is not diagnosed with Hereditary Angioedema (HAE) type 1/2
* The patient experienced ˂ 4 HAE attacks within last 12 month before enrolment in the study
* The participant is younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hereditary Angioedema type 1/2 patients
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-12 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Exploring the cleaved high-molecular weight kininogen (cHMWK) as a biomarker in HAE type 1/2 patients, as well as to study the differences between HAE type 1/2 patients without lanadelumab treatment versus patients on lanadelumab treatment. | 30 months
  Samples from HAE patients without lanadelumab treatment versus patients on lanadelumab treatment will be analyzed for cHMWK via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS).

SECONDARY OUTCOMES:
Studying cHMWK as a biomarker in HAE type 1/2 patients with edema attack, as well as to study the differences between HAE type 1/2 patients without lanadelumab treatment versus patients on lanadelumab treatment. | 30 months
  Samples from HAE patients without lanadelumab treatment versus patients on lanadelumab treatment collected before/during/after angioedema attacks will be analyzed for cHMWK via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS).

OTHER OUTCOMES:
Studying other metabolites as potential biomakers in HAE type 1/2 patients, as well as to study the differences between HAE type 1/2 patients without lanadelumab treatment versus patients on lanadelumab treatment. | 30 months
  All samples will be analyzed for potential biomarker candidates via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, MD, Study Chair — Centogene GmbH
Locations (7):
- Germany (7):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinik für Hals-Nasen-Ohrenheilkunde, Universitätsklinikum Düsseldorf,, Düsseldorf
  - Klinikum der Johann-Wolfgang-Goethe-Universität, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Universitäts-Hautklinik Leipzig, Leipzig
  - Hämophilie-Zentrum Rhein Main GmbH, Mörfelden-Walldorf
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No